CLINICAL TRIAL: NCT05498714
Title: Improved Bowel Cleansing Method for Colonoscopy Based on High Risk Population of Bowel Preparation#a Single-center,Endoscopist-blinded Randomized Controlled Trial
Brief Title: Improved Bowel Cleansing Method for Colonoscopy Based on High Risk Population of Bowel Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, ChenMingkai, Professor, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: WDRY2022-K082
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Bowel Preparation Before Colonoscopy
Keywords: Colonoscopy; Bowel Preparation; Polyethylene glycol; Compound Sodium Picosulfate; Lactulose
MeSH Terms: interventions — Lactulose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (Active Comparator): The dosing regimen of high-risk patients will be PEG combined with lactulose.
  Interventions: Drug: PEG+lactulose
- CSP+lactulose group (Experimental): The dosing regimen of high-risk patients will be CSP combined with lactulose.
  Interventions: Drug: CSP＋lactulose

INTERVENTIONS:
Drug: PEG+lactulose — On the day before colonoscopy , Patients took 50mL lactulose solution at 7:00 PM. And then Patients began to drink 1 L of PEG at 8:00 PM. On the day of the procedure, patients took 50 mL lactulose solution and the remaining 2 L of PEG 4-6 hours before colonoscopy.
  Other Names: PEG combined with lactulose
  Arms: the control group
Drug: CSP＋lactulose — On the day before colonoscopy , Patients took 50mL lactulose solution at 7:00 PM. And then Patients began to drink 150 mL of CSP at 8:00 PM ,followed by 2000ml of clarified liquid. On the day of the procedure, 4-6 hours before colonoscopy, patients took 50 mL lactulose solution and the remaining 150mL of CSP ,then followed by 750ml of clarified liquid .
  Other Names: CSP combined with lactulose
  Arms: CSP+lactulose group

SUMMARY:
The purpose of this study is to observe the difference in bowel preparation quality between compound sodium picosulfate#CSP combined with lactulose and polyethylene glycol electrolyte#PEG combined with lactulose in high-risk population.

DETAILED DESCRIPTION:
The quality of bowel preparation is crucial for colonoscopy. Some high-risk factors for inadequate bowel preparation have been identified , including age >70, previous colon surgery, constipation, diabetes, Parkinson's disease, history of stroke or spinal cord injury, prior history of inadequate bowel preparation, body mass index (BMI) >25, use of tricyclic antidepressant or narcotics. Patients were considered as high risk if they have any of the above factors.This is a single-center ,endoscopist-blinded study to compare the efficacy of CSP combined with lactulose and PEG combined with lactulose in bowel preparation. In colonoscopy procedures, endoscopists who were blinded to the intervention evaluated the overall quality of colonoscopy cleaning according to the Boston Bowel Preparation Scale. Patients' tolerance, defecation, adverse events and adenoma detection rate (ADR) were also evaluated.

ELIGIBILITY:
Inclusion Criteria:Adults undergoing colonoscopy who have at least one risk factor: age>70, previous colon surgery, constipation, diabetes, Parkinson's disease, history of stroke or spinal cord injury, prior history of inadequate bowel preparation, body mass index (BMI) >25, use of tricyclic antidepressant or narcotics.

Exclusion Criteria:

1. presence of any contraindications for colonoscopy (gastrointestinal obstruction or perforation,severe acute inflammatory bowel disease,toxic megacolon,severe heart failure,unable to swallow,severe heart failure,etc);
2. Patients with galactosemia;
3. hypersensitivity to any of the ingredients;
4. Pregnancy or lactation;
5. Use of lactulose,prokinetic agents or purgatives within 7 days;
6. Unwilling to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | during colonoscopy
  Cleanliness of the colon during colonoscopy will be evaluated by the Boston Bowel Preparation Scale which is a 4-point scoring system applied to each of 3 broad regions of the colon: the right side, the transverse section, and the left side. The total BBPS score ranged from 0 to 9. If total BostonBowel Preparation Score ≥6 with each segmental BBPS≥2, we regard it as adequate bowel preparation.

SECONDARY OUTCOMES:
Adenoma Detection Rate | 2 days
  Diagnosis was confirmed by histologic examination
Polyp Detection Rate | 2 days
  Diagnosis was confirmed by histologic examination
Rate of adverse events | 2 days
  adverse events, such as vomiting, nausea, headache, abdominal distention, abdominal pain.
Cecal intubation rate | during colonoscopy
  Colonoscopy reaches cecal region.
Cecal intubation time | during colonoscopy
  Colonoscopy reaches cecal region.
Withdrawal time | during colonoscopy
  The time from the cecum to the anus, but excluded time for biopsy performance or removal of polyps.
defecation frequency | 2 days
  Frequency of bowel movement.
patient satisfaction Assessment | 2 days
  Patients' satisfaction score for bowel preparation (3 points: completely tolerable and very satisfied; 2 points: nausea and other discomfort, but still tolerable and satisfactory; 1: unable to tolerate, not satisfied);
  And whether the patient is willing to use the bowel cleansing program for colonoscopy;

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, Ph.D & M.D, Study Director — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes